CLINICAL TRIAL: NCT01303497
Title: Phase II Study, Multicenter, Randomized, Stratified, Evaluating the Efficacity of Weekly Paclitaxel, With or Without Bevacizumab in the Treatment of Metastatic or Locally Advanced Angiosarcomas Not Accessible to Surgery Treatment.
Brief Title: Efficacity of Weekly Paclitaxel in Association or Not With Bevacizumab in Metastatic or Locally Advanced Angiosarcomas
Acronym: ANGIO-TAX+
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Collaborators: French Sarcoma Group (Other); Study Group of Bone Tumors (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANGIO-TAX-PLUS-0906
Record Dates: First submitted 2011-02-23; First posted 2011-02-24 (Estimated); Last update posted 2019-05-30 (Actual); Status verified 2017-01

CONDITIONS: Angiosarcoma
Keywords: Angiosarcoma; Paclitaxel; bevacizumab
MeSH Terms: conditions — Hemangiosarcoma | interventions — Paclitaxel; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A : Paclitaxel (Other): administration of paclitaxel drug during cycle of 28 days (6 cycles Max) + blood sample on day 1, 8, 15, 29 and 57
  Interventions: Drug: Paclitaxel
- Arm B : Paclitaxel + Bevacizumab (Other): administration of paclitaxel drug during per cycle of 28 days (6 cycles Max) + Bevacizumab every two weeks during paclitaxel cycles then every 3 weeks during P cycles until disease progression or inacceptable toxicity
  + blood sample on day 1, 8, 15, 29 and 57
  Interventions: Drug: Paclitaxel; Drug: Bevacizumab

INTERVENTIONS:
Drug: Paclitaxel — Day 1, 8 and 15 : Paclitaxel 90 mg/m², IV over 1h, during 6 cycles (1 cycle = 28 days)
  Other Names: Taxol
Drug: Bevacizumab — Bevacizumab until progression or inacceptable toxicity :
  * During the cycles of chemotherapy : Day 1 and D15 : 10 mg/kg,IV
  * After 6 cycles of chemotherapy : 15 mg/kg, IV
  Other Names: Avastin
  Arms: Arm B : Paclitaxel + Bevacizumab

SUMMARY:
Efficacity of Paclitaxel in association or not with Bevacizumab in treatment of angiosarcoma

DETAILED DESCRIPTION:
Randomization is stratified :

* angiosarcoma in irradiated region : yes / no
* visceral angiosarcoma : yes / no

All patient will received a maximum of 6 cycles of weekly Paclitaxel (Arm A and B) in association or not with Bevacizumab (ArmB).

1 cycle = 28 days Treatment by Bevacizumab is to continue beyond the 6th cycle, until disease progression or unacceptable toxicity

Arm A and B:

Day 1, D8 and D15 Paclitaxel : 90 mg/m², IV weekly with premedication

Arm B :

Day 1 and D15 Bevacizumab : 10 mg/kg and then, Bevacizumab : 15 mg/kg/3 weeks until disease progression or unacceptable toxicity

ELIGIBILITY:
Inclusion Criteria:

* Angiosarcoma histologically proven
* Metastatic or locally advanced and not accessible to surgery treatment
* Measurable tumor with at least 1 measurable lesion, according to RECIST
* For angiosarcoma in irradiated region, absence of clinical arguments of progression of the tumor prior treated by radiation
* At least 28 days since the previous treatment (systemic or major surgery)
* Performance Status (ECOG) ≤ 1
* Man or woman >= 18 years
* Polynuclear neutrophils >1500/mm3, platelets > 100 000/ mm3, Hemoglobin > 9.0 g/dl
* Total bilirubin ≤ 1.5 x USL, AST and ALT ≤ 2.5 x USL (or ≤ 5 if hepatic metastasis )
* Serum creatinin ≤ 1.5 x USL or clearance calculated > 50 ml/mn (Cockcroft formulae)
* Absence of hematuria on dipstick
* Proteinuria on dipstick <2+, if >2, the 24 hours proteinuria must be < 1g
* Albumin > 35 g/l and lymphocytes > 700/mm3 attesting a life expectancy > 3 months
* Normal cardiac function : LVEF ≥ 50%
* Normal coagulation test : INR ≤ 1.5 and TCA ≤ 1.5 x USL within 7 days before inclusion
* Systolic BP ≤ 150 mmHg and diastolic BP ≤ 100 mmHg
* Negative pregnancy test for women of reproductive potential(within 7 days before treatment start)
* Effective contraceptive methods for male and female (if applicable) during the period of treatment and until the 6 months after the last administration of Bevacizumab
* Adequate central veinous access
* Patient covered by government health insurance
* Informed consent form signed by the patient

Exclusion Criteria:

* Patients that have received more than 2 regimens of chemotherapy whatever the indication
* Kaposi's sarcoma, hemangio-endothelioma, hemangio-pericytoma (Malignant solitary fibrous tumor)
* Surgery (except the diagnostic biopsy) or radiotherapy within the past 4 weeks before inclusion, except antalgic radiotherapy
* Uncontrolled, active peptic ulcer,
* Other malignant evolutive tumor
* Previous thrombotic or hemorrhagic disorders
* Clinically significant cardiovascular disease (stroke within 6 months prior inclusion, unstable angina, heart failure, myocardial infarction, arrhythmia requiring treatment)
* Anticoagulant treatment for curative aim within 10 days before beginning of treatment (oral or parenteral administration), aspirin > 325 mg/day, or Plavix or a thrombolytic (thrombolytics for preventive use is permitted) or anti-platelet (dipyridamol, ticlopidine, clodiprogel, cilostazol)
* Chronic treatment(more than 15 days) by every AINS including aspirin > 325 mg/j
* Currently active bacterial or fungus infection (grade > 2 CTCAE v4.02)
* Known HIV1, HIV2, hepatitis B or hepatitis C infections
* Presence of known meningeal or brain metastasis
* Epilepsy requiring the use of anti-epileptic
* Previous organ transplant
* Peripheral stem cell transplantation within 4 months prior to inclusion in the study
* Using of drugs affecting the biological response, for example G-CSF, within the 3 weeks before inclusion
* Kidney dialysis patient
* Clinically significant neuropathy (grade> 2 CTCAE V4.02)
* Any circumstance that could jeopardise compliance or proper follow-up during the trial
* Pregnant or nursing women. Women should not breastfeed for at least 6 months after the last administration of Bevacizumab
* Constitutional or acquired coagulopathy
* Uncontrolled hypertension (SBP> 150 mmHg or DBP> 100 mmHg)
* Known hypersensitivity to paclitaxel or to one of its excipients (Cremophor EL, to Bevacizumab components, to products of Chinese hamster ovary cells (CHO) or other recombinant human or humanized antibodies
* Patients unable to undergo trail medical follow-up for geographical, social or psychological reasons
* Patient refusal of ambulatory care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2010-09-10 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2019-01-29 (Actual)

PRIMARY OUTCOMES:
Progression free rate after 6 months of treatment | after 6 months of treatment
  Stable disease, complete response and partial response according to RECIST 1.1

SECONDARY OUTCOMES:
Objective response at 3, 6, 9 months of treatment | at 3, 6, 9 months of treatment
  Stable disease, complete response and partial response according to RECIST 1.1
Median progression-free rate | an average time period of 1 year
  Median time for both cohort between :
  * date of inclusion
  * date of clinical or radiological progression
Global median survival | an average time period of 18 months
  Median time for both cohort between :
  * date of inclusion
  * date of death whatever the cause
Tolerance | during the study
  According to NCI-CTCAE v4.0
Correlation between efficacity and serum expression of anti angiogenic factors | Day 1, 8, 15, 29 and 57
  Blood samples at different times
Correlation between efficacity and beta-tubuline III expression in tissue | At baseline
  Paraffin blocks

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas PENEL, MD, PhD, Principal Investigator — Centre Oscar Lambret
Locations (13):
- France (13):
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Centre Val d'Aurelle, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - Centre René Gauducheau, Saint-Herblain
  - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lebellec L, Bertucci F, Tresch-Bruneel E, Ray-Coquard I, Le Cesne A, Bompas E, Blay JY, Italiano A, Mir O, Ryckewaert T, Toiron Y, Camoin L, Goncalves A, Penel N, Le Deley MC. Prognostic and predictive factors for angiosarcoma patients receiving paclitaxel once weekly plus or minus bevacizumab: an ancillary study derived from a randomized clinical trial. BMC Cancer. 2018 Oct 11;18(1):963. doi: 10.1186/s12885-018-4828-1. PMID 30305054